CLINICAL TRIAL: NCT06997146
Title: Identifying Biomarkers & Dysregulated Biological Pathways in Blood and Urine of Congenital Central Hypoventilation Syndrome (CCHS) Patients
Acronym: CCHSBiomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCHS Biomarkers
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Congenital Central Hypoventilation Syndrome (CCHS)
Keywords: CCHS; BIOMARKERS; POLYSOMNOGRAPHY; VENTILATORY SUPPORT; Metabolomic analyses
MeSH Terms: conditions — Congenital central hypoventilation syndrome | interventions — Blood Specimen Collection; Polysomnography; Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCHS Patient Group (Other): Participants in this arm are individuals diagnosed with Congenital Central Hypoventilation Syndrome (CCHS). They will undergo blood and urine sample collection at various timepoints during sleep and wakefulness. Additionally, they will undergo polysomnography to monitor sleep-related breathing patterns and to assess respiratory function during sleep. The focus is on analyzing biomarkers and dysregulated biological pathways associated with CCHS, and comparing them to matched healthy controls.
  Interventions: Biological: Blood and Urine Sampling; Device: Polysomnography; Other: lung function tests
- Matched Healthy Control Group (Other): Participants in this arm are healthy individuals who are matched for sex, age, origin, and BMI with the CCHS patients. They will undergo the same blood and urine sample collection at various timepoints during sleep and wakefulness, and will also undergo polysomnography to assess normal sleep patterns and respiratory function during sleep. This group serves as a comparison to understand the biomarkers and biological pathways in CCHS patients.
  Interventions: Biological: Blood and Urine Sampling; Device: Polysomnography; Other: lung function tests

INTERVENTIONS:
Biological: Blood and Urine Sampling — Collection of 10 mL of blood (separated into aliquots for RNA-seq and metabolomic analysis) and 5 mL of urine from participants at various timepoints during sleep and wakefulness. These samples will be used to analyze biomarkers and dysregulated biological pathways related to CCHS.
Device: Polysomnography — Participants will undergo polysomnography to assess sleep patterns and respiratory function during sleep. This will help evaluate any sleep-related breathing abnormalities in patients with CCHS and compare them with healthy controls.
Other: lung function tests — spirometry, ventilatory response to CO2

SUMMARY:
The CCHS study is a prospective, open-label, monocentric, interventional study with diagnostic and prognostic objectives, conducted in two phases. The first phase aims to identify biomarkers and dysregulated biological pathways in patients with Congenital Central Hypoventilation Syndrome (CCHS) by analyzing blood and urine samples of patients and matched healthy controls collected at multiple timepoints during sleep and wakefulness. In the second phase, these candidate biomarkers and pathways will be validated in a larger cohort of patients and matched healthy controls using targeted assays such as RT-PCR and mass spectrometry-based metabolomic analysis. The primary objective is to uncover molecular signatures that could explain disease mechanisms, while the secondary objective is to explore potential biomarkers and treatment targets that can improve spontaneous breathing and CO₂ responsiveness in CCHS patients. The underlying hypothesis is that multi-omics profiling of blood and urine can reveal actionable insights into the pathophysiology of CCHS and support the development of targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

CCHS patients :

1. Age 18 years old or older;
2. Carry a polyA expansion mutation in PHOX2B;
3. Receive nocturnal mechanical ventilation;
4. Patients that are under the care and treatment in the CCHS center: Hôpital Universitaire Pitié-Salpêtrière
5. Written informed consent from the patient
6. Affiliated to The French social security except patient on AME (state medical aid)

Control group :

1. Age 18 years old or older.
2. Healthy with no major medical illnesses in the past year (such as diabetes, cancer, pregnancy, lungs disease).
3. Matched for sex, age (+/- 3 years), origin and BMI category with a CCHS patient
4. Written informed consent of the control
5. Affiliated to The French social security except patient on AME (state medical aid)

Exclusion Criteria:

CCHS patients :

1. Age lower than 18 years old;
2. Pregnancy or breastfeeding
3. Patients with diaphragmatic (phrenic nerve) pacing;
4. Patients with late onset CCHS;
5. Patients that were diagnosed with a major medical illnesses/condition other than CCHS in the past year (such as diabetes, cancer, lungs disease, a sleep disorder, or pregnancy)
6. Patients that suffer from a sleep disorder such as insomnia, restless legs syndrome, nightmares
7. Patients who use medications that are likely to impair sleep structure
8. Individuals under guardianship, or permanently legally incompetent adults, under judicial protection, deprived of liberty, patients unable to express their consent.

Control group :

1. Age lower than 18 years old;
2. Pregnancy or breastfeeding
3. Controls that were diagnosed with a major medical illnesses/condition in the past year (such as diabetes, cancer, lungs disease, a sleep disorder, or pregnancy)
4. Controls that suffer from a sleep disorder such as insomnia, restless legs syndrome, nightmares
5. Controls who use medications that are likely to impair sleep structure.
6. Individuals under guardianship, or permanently legally incompetent adults, under judicial protection, deprived of liberty, patients unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Identification of dysregulated biological pathways and biomarkers in blood and urine of CCHS patients. | Day 0 to Month 37
  In the first phase of this study, candidate CCHS-related biomarkers and dysregulated pathways will be identified based on the analysis of the generated omics data. Candidate transcripts and metabolites that meet the criteria listed below will be further tested in the second targeted validation phase in an additional larger cohort of patients and matched controls. These will be sampled and analysed by specific tests (RT PCR or targeted metabolic analysis), that are relevant for each of the candidate transcripts and metabolites.
  The following criteria will be employed in the analyses of both phases:
  1. Significant alteration between patients and matched controls during sleep (and/or wakefulness).
  2. Significant alteration between sleep and wakefulness in controls.
  3. Significant alteration between sleep and wakefulness in patients.
  4. Significant alteration in the targeted validation phase, with a trend similar to the trend identified in phase I.

SECONDARY OUTCOMES:
Identify new CCHS prognostic biomarkers | Day 0 to Month 37
  New CCHS prognostic biomarkers will be identified by analyzing significant correlations between biomarker levels (such as RNA, metabolites, etc.) and performance on breathing tests in CCHS patients.
Discover new candidate treatment targets | Day 0 to Month 37
  The evaluation criteria for the identification and prioritization of new candidate treatment targets would include finding a solid scientific rational and defined and prioritized according to their parameters regarding pharmacodynamic-pharmacokinetic (PK/PD), ability to cross the blood brain barrier, drug developmental phase, regulatory status, intellectual property condition, and overall risk-benefit balance.
Identify relevant repurposed drugs/supplements | Day 0 to Month 37
  Relevant repurposed drugs/supplements will be defined and prioritized according to their parameters regarding pharmacodynamic-pharmacokinetic (PK/PD), ability to cross the blood brain barrier, drug developmental phase, regulatory status, intellectual property condition, and overall risk-benefit balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.